CLINICAL TRIAL: NCT04271228
Title: Use of Insulin Adjustment Device DreaMed Advisor Pro During Routine Clinical Use for Subjects With Diabetes Type 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC0525-19ctil
Record Dates: First submitted 2020-02-09; First posted 2020-02-17 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Type 1 Diabetes
Keywords: Decision Support System; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DreaMed Advisor Pro (Experimental): Using the DreaMed Advisor Pro as an advisory tool for Health Care Professionals during routine clinical use
  Interventions: Device: DreaMed Advisor Pro

INTERVENTIONS:
Device: DreaMed Advisor Pro — Using the DreaMed Advisor Pro as an advisory tool for Health Care Professionals during routine clinical use

SUMMARY:
The DreaMed Advisor Pro, is a software which automatically analyses treatment information, learns patient's needs and accordingly suggests adjustments in insulin dosing (FDA approved decision support system). The Advisor Pro uses information gathered from glucose monitoring (sensor readings or capillary blood glucose measurements), insulin dosing and meal data during daily routine home care. Following a 5 minute data collection and analysis, the algorithm learns and suggests pump-setting changes for optimization of glucose control. The algorithm is designed as an advisory tool for health care professionals and has three main components: First, data analysis report - a statistical analysis of the insulin pump and sensor data: insulin delivery, bolus-calculator rate of use, sensor glucose variables, hypoglycemic and hyperglycemic patterns. Second, recommendations, alert messages based on aforementioned data for example "pay attention- you skipped boluses", basal/bolus ratio is too high, bolus delivery compliance, glucose target recommendations and more. Third, a recommendation for new insulin pump settings: including basal intervals and rate, different carbohydrate ratio according to time of day, correction factor and insulin sensitivity time. The Advisor Pro can be used to optimize insulin pump setting during clinical visits, in-between visits or as part of virtual (telemedicine) visit. The objective of the proposed study is to evaluate the use of Advisor Pro by Health Care Providers for regular clinical visits and in between visits titration for adjustment of insulin pump settings. The study design is an open label, prospective, observational study that will include up to 100 participants with Type 1 Diabetes using insulin pumps and monitoring glucose levels by continuous glucose monitoring including flash glucose monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Documented Type 1 Diabetes for at least 1 year prior to study enrolment
* Subjects aged 6 - 65 years old
* HbA1c at inclusion ≤ 10%
* Subjects using Insulin pump therapy for at least 4 months
* Subjects using Insulin pump compatible with data transmission to the study Tidepool/Glooko Data Managment System (DMS) - Omnipod, Medtronic
* Subjects using Continuous Glucose Monitoring (CGM) System that is compatible with data transmission to the study Tidepool/Glooko DMS - Dexcom, Libre, Medtronic.
* Subjects willing to follow study instructions: Use CGM according to manufacture instructions, use the bolus-wizard feature of the insulin pump for every meal and correction boluses.
* Subjects have home PC or MAC connected to the internet.
* Subjects willing and able to sign a written informed consent form.

Exclusion Criteria:

* An episode of diabetic keto-acidosis within the month prior to study entry and/or severe hypoglycemia resulting in seizure or loss of consciousness in the month prior to enrolment.
* Concomitant diseases/ treatment that influence metabolic control or any significant diseases /conditions including psychiatric disorders and substance abuse that in the opinion of the investigator is likely to affect the subject's ability to complete the study or compromise patient's safety.
* Relevant severe organ disorders (diabetic nephropathy, diabetic retinopathy, diabetic foot syndrome) or any secondary disease or complication of diabetes mellitus, such as:

  1. Subject has unstable or rapidly progressive renal disease or is receiving dialysis
  2. Subject has active proliferative retinopathy
  3. Active gastroparesis
* Participation in any other interventional study
* Female subject who is pregnant or planning to become pregnant within the planned study duration
* Subject is in the "honeymoon" phase - i.e. less than 0.5 insulin units/kg per day.
* Known or suspected allergy to trial products
* Drug or alcohol abuse

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
HbA1c | Through study completion , an average of 1 year

SECONDARY OUTCOMES:
Percentage of glucose readings within target range of 70-180 mg/dl | Through study completion, an average of 1 year
Percentage of glucose sensor readings below 54 mg/dl | Through study completion, an average of 1 year
Percentage of glucose sensor readings above 250 mg/dl | Through study completion, an average of 1 year
Percentage of glucose sensor readings 70-54 mg/dl | Through study completion, an average of 1 year
Percentage of glucose sensor readings 180-250 mg/dl | Through study completion, an average of 1 year
Mean sensor glucose | Through study completion, an average of 1 year
Glucose variability | Through study completion, an average of 1 year
Total insulin dose | Through study completion, an average of 1 year
Total basal insulin dose | Through study completion, an average of 1 year
Total Bolus insulin dose | Through study completion, an average of 1 year
Total daily consumed carbohydrates | Through study completion, an average of 1 year

OTHER OUTCOMES:
Number of recommendations for changes in the treatment plan per patient | Through study completion, an average of 1 year
Number of physician overrides of advisor recommendations | Through study completion, an average of 1 year
Device satisfaction | at the end of the intervention period (1 year)
  Device satisfaction evaluated by Healthcare Professionals Survey containing 50 items, Device satisfaction evaluated by Healthcare Professionals Survey containing 50 items, 28 of them are on 5-point scale ranging from "strongly agree" to "strongly disagree", 10 items are "yes"/ "no" questions and 12 items are opened questions.
Frequency of home phone visits | Through study completion, an average of 1 year
Time required to review insulin pump and sensor data, make and send recommendations or length of visit | Through study completion, an average of 1 year
  will be measured by timer

CONTACTS AND LOCATIONS:
Overall Officials: Revital Nimri, MD, Principal Investigator — Schneider Children;s Medical Center
Locations (1):
- Schnider Children's Medical Center, Petah Tikva, Israel